CLINICAL TRIAL: NCT03150992
Title: A Feasibility Study of Elemental Diet as an Alternative to Parenteral Nutrition for Patients With Inoperable Malignant Bowel Obstruction
Brief Title: EDMONd - Elemental Diet in Bowel Obstruction
Acronym: EDMONd
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: University of Surrey (Other); Target Ovarian Cancer (Unknown)
Responsible Party: Principal Investigator, Agnieszka Michael, Consultant in Medical Oncology, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/LO/2079; 32895 (Other: NIHR Portfolio)
Record Dates: First submitted 2017-04-03; First posted 2017-05-12 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Ovarian Disease; Peritoneal Neoplasms; Peritoneal Diseases; Metastatic Ovarian Cancer; Primary Peritoneal Carcinoma; Abdominal Neoplasm; Bowel Obstruction
Keywords: Feasibility; Elemental Diet; Quality of life; Palliative; Nutrition; Ovarian; Peritoneal; Advanced; Metastatic; Bowel obstruction; Inoperable
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Diseases; Peritoneal Neoplasms; Peritoneal Diseases; Abdominal Neoplasms; Intestinal Obstruction; Neoplasm Metastasis | interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elemental 028 Extra Liquid (Experimental): All patients will be assessed and given an individual plan for Elemental Diet (ED) introduction. The actual amount of ED prescribed will depend on the tolerance and palatability and not nutritional status. The recommendation of a minimum of 2 cartons of ED will be drunk orally by patients, along with other clear fluids only. Following introduction of ED, patients will be discharged from hospital (if applicable) and followed up for 2 weeks. They will have a telephone follow-up assessment once a week for 2 weeks. All other assessments will follow the standard of care. During the follow-up patients will be assessed using the Memorial Symptom Assessment Scale (MSAS) and will be asked to complete a nutritional diary every day and a quality of life questionnaire at several time points.
  Interventions: Dietary Supplement: Elemental 028 Extra Liquid

INTERVENTIONS:
Dietary Supplement: Elemental 028 Extra Liquid — A nutritionally complete, liquid elemental diet consisting of a mixture of essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals, trace elements and flavourings with sugars & sweeteners.
  Other Names: Elemental Diet

SUMMARY:
A feasibility study to provide 'proof of concept' of Elemental Diet (ED) as an acceptable/ useful feeding option for patient with inoperable malignant bowel obstruction and to examine the impact of ED on quality of life

DETAILED DESCRIPTION:
The aim of this study is to determine whether Elemental Diet (a type of drink that contains an elemental protein source known as amino acids) can be tolerated by patients with inoperable bowel blockage who can no longer eat and are only able to swallow small amount of fluid. The objective is to find out whether elemental diet (ED) can be used as an acceptable nutrition and whether it improves the quality of life. Bowel blockage is a common complication in patients with ovarian cancer. Unfortunately when the cancer is advanced, this blockage can occur in many parts of the bowel therefore surgery is not possible. Every year in the UK some publications report the rate as high as 50% . One way to feed patients with bowel blockage is through the veins; this is known as parenteral nutrition (PN) however PN is rarely used in United Kingdom. Patients with malignant bowel blockage are often able to swallow small amounts of liquid but if they have no PN they are only able to survive for 2-3 weeks and the psychological as well as physical impact on patients and the family are very distressing. ED is a type of a drink which contains an elemental protein source known as amino acids. ED drinks are almost totally absorbed in the upper part of the bowel and therefore could be absorbed even in patients who have bowel blockage which usually develops lower down in the gut. If this study is successful and proves that ED can be tolerated and provide nutrition to patients with inoperable bowel blockage it will be a big step towards improving the quality of life at the final stage of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed inoperable bowel obstruction due to disseminated malignancy
* Ability to tolerate 500ml of liquid
* Capacity to give informed consent

Exclusion Criteria:

* Bowel obstruction that can be managed with surgical intervention
* Complete bowel obstruction and inability to tolerate small amount of liquid

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Taste acceptability of ED | Two weeks
  Taste of at least one flavor of ED graded as 2 out of 5 by patient on nutritional diary taste acceptability scale (1=I really like the taste, 2=I like the taste, 3=The taste is acceptable, 4=I do not like the taste but can drink it, 5=I do not like the taste and cannot drink it).
Change in incidence of vomiting | Two weeks
  No deterioration in incidence of vomiting as measured on MSAS scale. Grading 1 (occurring rarely) or 2 (occurring occasionally) is acceptable. Deterioration considered as change to 3 (occurring frequently) or 4 (occurring almost constantly).
Change in incidence of pain | Two weeks
  No deterioration in incidence of abdominal pain as measured on MSAS scale. Grading 1 (occurring rarely) or 2 (occurring occasionally) is acceptable. Deterioration considered as change to 3 (occurring frequently) or 4 (occurring almost constantly).

SECONDARY OUTCOMES:
The number of patients who can tolerate ED following presentation with IBO and can subsequently be treated with palliative chemotherapy | Two weeks
  Measured by reviewing hospital case notes
Number of patients alive at the end of the study | Up to two years
  Measured by reviewing hospital case notes
Health related quality of life | Two weeks
  Measured on EORTC-QLQ-C30
Nutritional intake | Two weeks
  Measured by number of cartons taken by patient in 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Michael, MBBS PhD, Principal Investigator — Royal Surrey County Hospital, University of Surrey
Locations (1):
- Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No